CLINICAL TRIAL: NCT05679193
Title: Perioperative Propranolol in Robotic Assisted Laparoscopic Prostatectomy- A Feasibility Study of Propranolol to Target Perioperative Stress Induced Cancer Progression
Brief Title: Perioperative Propranolol During Prostatectomy to Decrease Cancer Recurrence
Acronym: PeP-RALP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Ivar, Ragna og Morten Holes legat til fremme av kreftforskningen i Norge (Unknown); Fondsstiftelsen ved Oslo Universitetssykehus (Unknown)
Responsible Party: Principal Investigator, Shivanthe Sivanesan, Urologist and General Surgeon, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 488466
Record Dates: First submitted 2022-12-12; First posted 2023-01-10 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: parallel-group, phase 2, double-blind, 2-arm study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol (Experimental): Participants will receive Propranolol capsule for a period of 22-28 days, low dose (1 capsule/20mg propranolol twice daily) treatment the first- and last- three days of the treatment period. Higher dose (2 capsules/40mg propranolol twice daily) for the rest of the treatment period.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Participants will receive Propranolol capsule for a period of 22-28 days, low dose (1 capsule twice daily) treatment the first- and last- three days of the treatment period. Higher dose (2 capsules twice daily) for the rest of the treatment period.
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol capsules 20mg taken orally.
  Day: 1-3:
  20mg twice daily
  Day: 4-19 (25 , In cases of delayed RALP an extension of up to 6 days is allowed.in cases of delayed surgery).
  2x 20mg twice daily
  Day 20-22 20mg twice daily
  Other Names: Pranolol

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a larger randomized controlled trial to assess the efficacy of perioperative propranolol capsules compared with placebo capsules in decreasing recurrence of prostate cancer (PCa) after robotic assisted laparoscopic prostatectomy (RALP) in participants with intermediate to high-risk for prostate cancer recurrence.

DETAILED DESCRIPTION:
PCa is the most commonly diagnosed cancer in Norway (2020) and RALP is the most frequent curative treatment offered to men with non-metastatic PCa. Biochemical recurrence (BCR) is estimated to occur to 40% of patients with EAU IR and HR PCa. Attempts to combat the high recurrence rates after RALP with neoadjuvant treatment, aiming to reduce the local tumor burden and treat possible micrometastasis, has of yet not proven beneficial.

The prostate is highly innervated and recent evidence has shown the importance of nerves in the development and progression of PCa. The action of particularly adrenergic nerves, in sum lead to a pro-cancerous and metastatic state by influencing key hallmarks of cancer like apoptosis resistance, angiogenesis, immune suppression, invasiveness and metastasis.

Perioperative stress caused by the cancer surgery, in this case RALP, has been found to promote cancer progression and recurrence both by enhancing growth of preexisting residual tumor/micrometastasis and facilitating formation of new metastasis. The surgical stress response cause a catecholamine-induced cancer progression where β2-adrenergic receptor (ADRB2) have a key role.

Our newly published pharma co-epidemiologic study indicate perioperative stress can be targeted by a non-selective ß-blocker (nsBB) like propranolol [1]. RCTs have found perioperative administration of propranolol alone, or in conjunction with COX-2 inhibition, to be safe and to reduce biomarkers associated with poor prognosis compared with the control group receiving placebo medication in patients undergoing radical surgery for breast-, ovarian- and colorectal cancer [2-7}.

The result of our register study, together with existing evidence of an effect of propranolol/nsBBs, provides foundation for PeP-RALP, a pilot study to establish the recruitment- and infrastructure feasibility of a double-blinded, placebo controlled RCT. The results of this pilot study will be used to investigate the feasibility of a formal larger RCT aiming to assess efficacy of perioperative propranolol to reduce PCa recurrence and progression after RALP.

ELIGIBILITY:
Inclusion Criteria:

* European Association of Urology Intermediate- and High Risk for Biochemical recurrence and planned for curative RALP
* ECOG Performance Status 0-1

Exclusion Criteria:

Medical Conditions

1. Sick sinus syndrome
2. Atrioventricular (AV) block grade 2 and 3
3. Recent (3 months) myocardial infarction
4. Known unstable- or vasospastic- angina
5. Heart failure (New York Heart Association [NYHA] > 2)
6. Symptomatic peripheral vascular disease (e.g. intermittent claudication)
7. Known pulmonary hypertension
8. Known carotid artery stenosis or recent (3 months) stroke
9. Bronchial asthma or other chronic obstructive pulmonary disease (COPD)
10. Kidney failure (estimated Glomerular filtration rate [eGFR]<50)
11. Liver failure (cirrhosis, jaundice, signs of hepatic decompression)
12. Unregulated diabetes mellitus
13. Untreated thyroid disorder
14. Depressive episode within last 6 months (within last 12 months if major depressive episode)
15. Known drug allergy against propranolol or excipients
16. Any medical conditions considered to prohibit Propranolol use as judged by the treating physician (including frailty).
17. Participants with known substance- or alcohol-abuse

    Prior/Concomitant Therapy
18. Recent (<3 month) use of systemic beta-blockers prior to screening.
19. Patients receiving non-dihydropyridine calcium channel blocking agents (eg diltiazem, verapamil)
20. Patients receiving anti-arrhythmic agents (e.g. amiodarone, sotalol, digoxin, verapamil, flecainide)
21. Patients receiving digoxin, rizatriptan, hydralazine, fluvoksamin, or fluoksetin
22. Patients using daily anxiolytics (e.g. benzodiazepines), alpha-receptor adrenergic agonists (e.g. clonidine)
23. Recommendations in the Summary of Product Characteristics for propranolol regarding concomitant use of other medications will be adhered to.

    Diagnostic assessments
24. Sinus bradycardia (<60 beats/minute)
25. Resting blood pressure <110/60mmHg OR hypertension BP >160/100
26. AV-block 2 or 3 on ECG

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
The feasibility of conducting a formal larger RCT to compare the efficacy of propranolol vs placebo to decrease PCa recurrence following RALP. | The total duration of study participation from screening to end of follow-up is 50-102 days per participant. The primary outcome will be assessed when inclusion is completed, or if inclusion is not completed within 12 months.
  Numbers of eligible participants needed to screen to include 40 patients in the study, reported as % of eligible participants that subsequently were included in the study.
  Compliance of study intervention (defined as >80% of doses taken). Reported as % of participants compliant to the study intervention before RALP and % of participants compliant to the study intervention after RALP.

SECONDARY OUTCOMES:
Safety and tolerability of PeP-RALP intervention | 9 weeks
  Safety:
  Proportion (%) of patients experiencing treatment related clinical significant hypotension and/or bradycardia.
  Adverse events of PeP-RALP medication as assessed by CTCAE v5.0.
  Tolerability:
  Proportion (%) of patients tolerating daily dose of 80mg propranolol.
Determine the effect of RALP on catecholamine levels | Up to 5 weeks
  Changes in catecholamine levels in the perioperative period.
Determine the bioavailability of propranolol | Up to 5 weeks
  Serum levels of propranolol pre-operatively and at end of PeP-RALP medication.
Determine the effect of preoperative propranolol treatment on the serum level of PSA | 7-14 days
  Changes in PSA levels after 7-14 days of PeP-RALP medication.
To determine the effect of propranolol on post-operative biochemical failure | Up to 9 weeks
  Proportion of patients with serum PSA levels above 0.1 ng/ml at 6 weeks post-RALP.
Intraoperative anesthesiological and surgical challenges Surgical complications in PeP RALP patients | 1 day
  Anesthesiological challenges are assed by:
  Proportion of patients (%) in each intervention group requiring vasopressors to maintain an acceptable mean arterial pressure (MAP >60mmhg). Amount of vasopressor needed.
  Surgical challenges are assed by:
  The surgical procedure time (minutes) and estimated intraoperative blood loss (milliliters).
Surgical complications | Up to 9 weeks
  Frequence (n=) and severity of surgical complications as classified by the Clavian-Dindo classification.

OTHER OUTCOMES:
Change in perceived distress during the study. | Up to 9 weeks
  Investigate alterations in perioperative perceived distress, assessed by Hospital Anxiety and Depression Scale (HADS)
Immunohistochemistry and Image mass cytometry of tumor to assess for differences between treatment arms. Flow cytometry to assess of periferal blood to assess for differences between treatment arms. | Up to 9 weeks
  Immunohistochemistry and image mass cytometry to assess for differences between treatment arms in intra-tumor immune cell infiltration.
  Flow cytometry to assess differences between treament arms in systemic immune cell acitivity.
Difference in prognostic markers (e.g. Decipher GRID transcriptome analysis) between treatment arms. Identify predictive biomarkers for propranolol responsiveness (e.g. Decipher GRID transcriptome analysis) | up to 1 year
  Determine the effect of pre-operative propranolol treatment on prognostic markers and assess for predictive biomarkers. Identify predictive biomarkers for propranolol responsiveness.
Differences between intervention arms with regard to intraoperative alterations in cerebral autoregulation and intracranial pressure, measured by transcranial doppler (TCD) floe velocity. | up to 1 year
  Intraoperative alterations in cerebral autoregulation and intracranial pressure by Transcranial Doppler flow velocity measurement of the middle cerebral artery.

CONTACTS AND LOCATIONS:
Overall Officials: Shivanthe Sivanesan, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital The Norwegian Radium Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
IPD that underlie the results reported in a published articles based on this study, after deidentification (text, tables, figures, and appendices)

REFERENCES:
- [Background] Sivanesan S, Tasken KA, Grytli HH. Association of beta-Blocker Use at Time of Radical Prostatectomy With Rate of Treatment for Prostate Cancer Recurrence. JAMA Netw Open. 2022 Jan 4;5(1):e2145230. doi: 10.1001/jamanetworkopen.2021.45230. PMID 35080602
- [Background] Zhou L, Li Y, Li X, Chen G, Liang H, Wu Y, Tong J, Ouyang W. Propranolol Attenuates Surgical Stress-Induced Elevation of the Regulatory T Cell Response in Patients Undergoing Radical Mastectomy. J Immunol. 2016 Apr 15;196(8):3460-9. doi: 10.4049/jimmunol.1501677. Epub 2016 Mar 11. PMID 26969754
- [Background] Hiller JG, Cole SW, Crone EM, Byrne DJ, Shackleford DM, Pang JB, Henderson MA, Nightingale SS, Ho KM, Myles PS, Fox S, Riedel B, Sloan EK. Preoperative beta-Blockade with Propranolol Reduces Biomarkers of Metastasis in Breast Cancer: A Phase II Randomized Trial. Clin Cancer Res. 2020 Apr 15;26(8):1803-1811. doi: 10.1158/1078-0432.CCR-19-2641. Epub 2019 Nov 21. PMID 31754048
- [Background] Shaashua L, Shabat-Simon M, Haldar R, Matzner P, Zmora O, Shabtai M, Sharon E, Allweis T, Barshack I, Hayman L, Arevalo J, Ma J, Horowitz M, Cole S, Ben-Eliyahu S. Perioperative COX-2 and beta-Adrenergic Blockade Improves Metastatic Biomarkers in Breast Cancer Patients in a Phase-II Randomized Trial. Clin Cancer Res. 2017 Aug 15;23(16):4651-4661. doi: 10.1158/1078-0432.CCR-17-0152. Epub 2017 May 10. PMID 28490464
- [Background] Haldar R, Shaashua L, Lavon H, Lyons YA, Zmora O, Sharon E, Birnbaum Y, Allweis T, Sood AK, Barshack I, Cole S, Ben-Eliyahu S. Perioperative inhibition of beta-adrenergic and COX2 signaling in a clinical trial in breast cancer patients improves tumor Ki-67 expression, serum cytokine levels, and PBMCs transcriptome. Brain Behav Immun. 2018 Oct;73:294-309. doi: 10.1016/j.bbi.2018.05.014. Epub 2018 May 22. PMID 29800703
- [Background] Jang HI, Lim SH, Lee YY, Kim TJ, Choi CH, Lee JW, Kim BG, Bae DS. Perioperative administration of propranolol to women undergoing ovarian cancer surgery: A pilot study. Obstet Gynecol Sci. 2017 Mar;60(2):170-177. doi: 10.5468/ogs.2017.60.2.170. Epub 2017 Mar 16. PMID 28344958
- [Background] Haldar R, Ricon-Becker I, Radin A, Gutman M, Cole SW, Zmora O, Ben-Eliyahu S. Perioperative COX2 and beta-adrenergic blockade improves biomarkers of tumor metastasis, immunity, and inflammation in colorectal cancer: A randomized controlled trial. Cancer. 2020 Sep 1;126(17):3991-4001. doi: 10.1002/cncr.32950. Epub 2020 Jun 13. PMID 32533792